CLINICAL TRIAL: NCT01459354
Title: The Effects of Bimanual Laryngoscopy on Post-Operative Sore Throat in Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DMR100-IRB-146
Record Dates: First submitted 2011-10-23; First posted 2011-10-25 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Postoperative Sorethroat; Bimanual Laryngoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- post, bimanual laryngoscopy, POGO score: one control, one study group

SUMMARY:
Post-operative sore throat, cough, and hoarseness of voice are common, uncomfortable, distressing sequelae after tracheal intubation. It was postulated that these effects are because of irritation and inflammation of the airway. Bimanual laryngoscopy is known to improve visual field during intubation. This procedure might reduce laryngeal trauma during intubation and therefore reduce the incidence or degree of post-operative sore throat. This is the first prospective, double-blinded, controlled study, which is focused on the effects of bimanual laryngoscopy on first 24-houred post-operative sore throat (POST).

ELIGIBILITY:
Inclusion Criteria:

1. ASA I or II
2. 20-70 y/o
3. GAET for A. Breast op B. GYN op C. Upper/lower extremities op D. Ophthalmology op E. GU op F. minor surgery

Exclusion Criteria:

1. emergency surgery
2. head and neck surgery
3. recent URI symptom in last one weeks with medication
4. post op PCA use
5. on NG/OG
6. perioperative bucking

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20-70 yrs patient receive elective surgery with general anesthesia without position change or any influence on sorethroat
Sampling Method: Probability Sample
Enrollment: 490 (Estimated)
Dates: Start 2011-08

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan ROC, Taiwan